CLINICAL TRIAL: NCT00142103
Title: CPG10101 Combination Therapy For The Treatment Of Hepatitis C: A Phase 1b Open Label Randomized Trial Of CPG10101 Alone, With Interferon, Ribavirin, Or Interferon And Ribavirin In The Treatment Of Relapsed Hepatitis C Virus (HCV) Subjects
Brief Title: CPG10101 Combination Therapy For The Treatment Of Hepatitis C In Relapsed Hepatitis C Virus (HCV) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1211001; CPG10101-003
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Hepatitis, Chronic Active
Keywords: Hepatitis c virus; HCV; Liver
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- CPG10101 (Experimental)
  Interventions: Drug: CPG10101
- CPG10101 + pegylated interferon (Experimental)
  Interventions: Drug: CPG10101
- CPG10101 + ribavirin (Experimental)
  Interventions: Drug: CPG10101
- CPG10101 + pegylated interferon + ribavirin (Experimental)
  Interventions: Drug: CPG10101
- Pegylated inteferon + ribavirin (Active Comparator)
  Interventions: Drug: Control
- CPG10101 + pegylated interferon + ribavirin (rollover) (Experimental)
  Interventions: Drug: CPG10101

INTERVENTIONS:
Drug: CPG10101 — CPG10101 subcutaneous, 0.20mg/kg, weekly, 12wks
  Arms: CPG10101
Drug: CPG10101 — CPG10101, subcutaneous, 0.20mg/kg, weekly, 12wks Pegylated Interferon alfa-2b, subcutaneous, 1.5ug/kg, weekly, 12wks
  Arms: CPG10101 + pegylated interferon
Drug: CPG10101 — CPG10101, subcutaneous, 0.20mg/kg, weekly, 12wks Ribavirin, oral, 800-1400mg, daily, 12wks
  Arms: CPG10101 + ribavirin
Drug: CPG10101 — CPG10101, subcutaneous, 0.20mg/kg, weekly, 12wks Pegylated Interferon alfa-2b, subcutaneous, 1.5ug/kg, weekly, 12wks Ribavirin, oral, 800-1400mg (weight-based), daily, 12wks
  Arms: CPG10101 + pegylated interferon + ribavirin
Drug: Control — Pegylated Interferon alfa-2b, subcutaneous, 1.5ug/kg, weekly, 12wks Ribavirin, oral, 800-1400mg (weight-based), daily, 12wks
  Arms: Pegylated inteferon + ribavirin
Drug: CPG10101 — CPG10101, subcutaneous, 0.20mg/kg, weekly, 12wks Pegylated Interferon alfa-2b, subcutaneous, 1.5ug/kg, weekly, 12wks Ribavirin, oral, 800-1400mg (weight-based), daily, 12wks
  Arms: CPG10101 + pegylated interferon + ribavirin (rollover)

SUMMARY:
1. To characterize the tolerability profile of subcutaneous (SC) CPG 10101 alone, with pegylated interferon, ribavirin or both pegylated interferon and ribavirin when administered weekly for twelve weeks in relapsed HCV positive subjects.
2. To assess the effect of subcutaneous (SC) CPG 10101 alone, with pegylated interferon, ribavirin or both pegylated interferon and ribavirin on serum Hepatitis C Virus (HCV) RNA concentrations

ELIGIBILITY:
Inclusion Criteria:

HCV positive subjects documented by serum HCV RNA concentration greater than 1000 IU/mL within 21 days of first study treatment.

Receipt of adequate pegylated IFN plus RVN based therapy for a minimum of 24 weeks (pegylated interferon doses of > 180 μg weekly or > 1.0 μg/kg pegylated interferon weekly and at least 800 mg RVN daily) resulting in undetectable HCV RNA concentrations while on treatment with subsequent relapse (HCV RNA concentration detected) within six months of stopping therapy.

HCV genotype 1. Adults, 18 + years old. Written Informed Consent. Liver biopsy documenting changes of Hepatitis C within 5 years of the first dose of study drug.

Adequate bone marrow, liver, and renal function demonstrated by:

* hemoglobin > 12 g/dL for females and > 13 g/dL for males
* WBC > 3,000/mm3
* Neutrophils > 1,500/mm3
* Platelets > 80,000/mm3
* Total bilirubin < 1.6 mg/dL.
* Direct bilirubin < 1.5 upper limit of normal. If indirect bilirubin is elevated, Gilbert's disease must be documented in chart and substantiated.
* Albumin within normal limits (per central laboratory)
* Serum creatinine < upper limit normal per central laboratory or calculated creatinine clearance > 100 mL/min (by Cockroft-Gault formula).

Negative pregnancy test in women of child bearing potential Females of childbearing potential and males who have partners of childbearing potential must use two forms of effective contraception during treatment and during the 6 months after treatment has been concluded.

Exclusion Criteria:

Treatment with IFN based therapies and/or antiviral therapies within 90 days of the first dose of study drug.

Child-Pugh Class B or C. History of psychiatric conditions including, but not limited to, psychosis, suicidal ideations, or major depression. Subjects with mild to moderate depression in the past who have a normal to mild Beck Depression Inventory Score and no prior history of suicidal gestures or attempts may be enrolled if, in the Investigator's opinion, they are suitable for treatment.

Significant cardiovascular disease (e.g., NYHA class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).

History of immunodeficiency, autoimmune disease, autoimmune hepatitis, allogeneic transplant, or pre-existing autoimmune or antibody-mediated disease including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia.

Other serious medical conditions including, but not limited to:

* HIV-1,
* Hepatitis B (positive HBsAg),
* Cancer,
* Pregnant, partners of pregnant women, or nursing women, and/or
* Alcohol or drug misuse within 90 days of screening Use of immunosuppressive doses of steroids or any antimetabolite therapies within 3 months of entry into the study (inhaled and topical corticosteroids are permitted).

Receipt of any vaccine or immunoglobulin within 30 days before the first dose of study drug Prior administration of oligodeoxynucleotides (including study medication CPG 10101), ribozymes, or any known allergy to CPG 10101, interferon, ribavirin or their excipients Receipt of any investigational drug therapy within 30 days before the first dose of study drug Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs, clinical and laboratory parameters, physical exam, ECG | 16wks

SECONDARY OUTCOMES:
Serum HCV RNA concentrations: Serum HCV concentrations over time to baseline | 12wks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1211001&StudyName=CPG10101%20Combination%20Therapy%20For%20The%20Treatment%20Of%20Hepatitis%20C%20In%20Relapsed%20HCV%20Subjects